CLINICAL TRIAL: NCT05887258
Title: Randomized Clinical Trial to Compare the Efficacy of Opioid-free Vs Traditional Balanced Anesthesia in Laparoscopic Colorectal Surgery
Brief Title: Opioid-free Vs Traditional Balanced Anesthesia in Laparoscopic Colorectal Surgery
Acronym: OFA_GAL_21
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Unai Ortega Mera (Other)
Collaborators: Osakidetza (Other)
Responsible Party: Sponsor-Investigator, Unai Ortega Mera, Principal Investigator, Osakidetza
Organization: Osakidetza (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-003245-38
Record Dates: First submitted 2023-04-16; First posted 2023-06-02 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid free anesthesia (OFA) (Experimental): This arm is administered by the anesthesiologist in charge of the operating room.
  It is composed by Dexmedetomidine (Dexdor), Lidocaine, Magnesium Sulfate and ketamine (Ketolar).
  Interventions: Drug: Opioid free anesthesia
- Opioid based Anesthesia (OA) (Active Comparator): This arm is administered by the anesthesiologist in charge of the operating room.
  This arm is composed of Remifentanil hydrochloride and postoperative rescue analgesia will be morphine.
  Interventions: Drug: Opioid based Anesthesia

INTERVENTIONS:
Drug: Opioid free anesthesia — It administers a combination of drugs to replace the opioid derivatives. Among them, we will use lidocaine, ketamine, dexmetomidine, and magnesium sulfate in continuous infusion adjusted to the patient's weight during surgery.
  Other Names: OFA
  Arms: Opioid free anesthesia (OFA)
Drug: Opioid based Anesthesia — administer anesthesia based on opioids such as fentanyl and/or morphine to guarantee analgesia during the surgical intervention.
  Other Names: Traditional anesthesia
  Arms: Opioid based Anesthesia (OA)

SUMMARY:
The goal of this clinical trial is to compare opioid free anesthesia versus opioid anesthesia in patients undergo laparoscopic colorectal surgery. The main question it aims to answer is assess the efficacy of opioid-free anaesthesia respect to postoperative pain control in patients undergoing a laparoscopic colorectal surgery.

Participants will answer a questionnaire during the first 3 days of admission, assessing pain through the visual analog scale (VAS).

The researchers will compare the consumption of opiates during the postoperative period in the opioid-free anesthesia group.

DETAILED DESCRIPTION:
The objective of the study is to know the efficacy of OFA in laparoscopic colorectal surgery. The consumption of opiates will be evaluated according to the VAS scale, defining non-tolerable pain greater than 5. The number of rescues required, the time elapsed until the first rescue and the total consumption of opiates administered will be evaluated.

Other variables that will be evaluated will be safety variables defined as intraoperative complications that require immediate action by the anesthesiologist, interruption of the procedure, or conversion to open surgery.

Other variables evaluated will be postoperative complications:

* Postoperative hypoxemia.
* Incidence of postoperative nausea and vomiting (PONV).
* Postoperative ileus.
* surgical complications.
* medical complications

ELIGIBILITY:
Inclusion Criteria:

( - ) Patients older than or equal to 18 years.

(-) Patients scheduled for laparoscopic colorectal surgery.

(-) Patients with physical status classification (ASA) I-III.

(- ) Patients who have signed the informed consent of the clinical trial

Exclusion Criteria:

(-) Pregnant or lactating patients.

(-)Patients with allergy to any of the drugs or excipients used in the study

(-) Emergency laparoscopic colorectal surgery

(-) Patients with AV block, intraventricular block, or sinus block

(-) Adam-Stokes syndrome.

(-) Patient on chronic beta-blocker treatment with HR < 50 bpm

(-) Patient with ejection fraction < 40% known

(-) Epilepsy.

(-) Surgery converted to open surgery

(-) Legally disabled patient

(-) Patients with physical status classification (ASA) IV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Pain control | 3 days
  milligrams of opioids required postoperatively during the first 3 of admission

SECONDARY OUTCOMES:
VNS score | 3 days
  Pain measured through the visual analogue scale (VAS) during the first 3 days of admission
morphine rescues | 7 days
  Number of opiate rescues required during the postoperative period

OTHER OUTCOMES:
intraoperative Security | 1 day
  Presentation of complications during the surgical intervention defined as a situation that requires immediate action by the anesthetist and lasts more than 30 minutes, the interruption of the operation and/or conversion to open surgery.
postoperative security | 3 day
  Operative hypoxemia defined as oxygen saturation by pulseoximetry less than 90% Incidence of Postoperative Nausea and Vomiting (PONV) during de first 3 days Postoperative ileus defined as the absence of bowel movements during the first 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Unai Ortega, MD, Principal Investigator — Osakidetza
Locations (1):
- Hospital de Galdakao, Galdakao, Vizcaya, Spain

IPD SHARING:
Plan to Share IPD: No